CLINICAL TRIAL: NCT07199972
Title: Trajectory of COVID-Related Tinnitus Over the Pandemic Timeline
Brief Title: COVID-Related Tinnitus Timeline
Acronym: TinCovTime
Status: Completed | Type: Observational
Sponsor: Faculdade de Medicina de Valenca (Other)
Responsible Party: Principal Investigator, Ricardo Rodrigues Figueiredo, MD,MSc,PhD, Faculdade de Medicina de Valenca
Other Study IDs: TinCOVID
Record Dates: First submitted 2025-09-28; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Hearing Disorders; COVID-19 Pandemic
Keywords: covid-19; tinnitus
MeSH Terms: conditions — Hearing Disorders; COVID-19; Tinnitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 is a respiratory disease caused by the coronavirus SARS-CoV-2, for which the first cases were reported in China, by December 2019. Previous studies reported cases of tinnitus following COVID infection, most of them mild and with similar characteristics to other forms of tinnitus. Our aim is to further explore the relationship between COVID-19 and tinnitus. For this purpose we analyzed people in the city of Volta Redonda, Brazil after a COVID-19 infection. In detail we compared those with new onset tinnitus during or after COVID-19 with those without tinnitus and those with tinnitus onset before the COVID-19 infection. Moreover we analyzed the prevalence of post-COVID tinnitus along the pandemic timeline, from 2020 to 2024.

DETAILED DESCRIPTION:
Two-hundred and thirty three patients over 18 years old and previously diagnosed with COVID-19 confirmed by either a RT-PCR, antibodies or antigens test were included. Patients were subdivided in three groups: no tinnitus (NT), tinnitus that already existed before COVID-19 (chronic tinnitus, CT) and tinnitus that arose during or after COVID-19 (post-COVID-19 tinnitus, PCT). Data concerning COVID-19 symptoms, drugs prescribed for COVID-19, tinnitus characteristics, comorbidities and other otological symptoms were collected. Tinnitus assessment included pure tone audiograms, the Tinnitus Handicap Inventory (THI), visual-analog scales (VAS) for loudness and distress as well as the hospital anxiety and depression scale (HADS). Patients with CT were additionally asked whether their tinnitus worsened after their COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

* previous COVID-19 infection

Exclusion Criteria:

* < 18 yo
* not willing to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who had a previous COVID-19 infection
Sampling Method: Non-Probability Sample
Enrollment: 233 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Trajectory of COVID-Related Tinnitus Over the Pandemic Timeline | February 2023 - November 2024
  Post-COVID tinnitus x No tinnitus x chronic tinnitus

CONTACTS AND LOCATIONS:
Overall Officials: Norma O Penido, MD,PhD, Study Chair — Universidade Federal de São Paulo
Locations (1):
- OTOSUL, Otorrinolaringologia Sul-Fluminense, Volta Redonda, Rio de Janeiro, Brazil